CLINICAL TRIAL: NCT01536769
Title: Intestinal and Nasal Microbiota of Patients With Idiopathic Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Jorvi Hospital (Unknown); Hyvinkää Hospital (Other); Peijas Hospital (Unknown); University of Helsinki (Other)
Responsible Party: Principal Investigator, Filip Scheperjans, Neurologist, Helsinki University Central Hospital
Other Study IDs: 86/2011
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Parkinson's Disease
Keywords: Metagenomic analysis; Microbiota
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Nasal and oral bacterial swabs and stool samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinson patients: Parkinson patients, symptom onset > 50 years of age, non-smoker, no relevant gastrointestinal or ENT diseases
- Control subjects: No parkinsonism, age and gender matched to PD subjects, non-smoker, no relevant gastrointestinal or ENT diseases

SUMMARY:
The cause of Parkinson's disease (PD) is unknown and a reliable biomarker to identify PD patients as early as possible is urgently needed. Nerve cells near the nose and in the gut become first affected in PD and patients frequently suffer from loss of smell and constipation. The nose and gut harbor very high amounts of bacteria that influence our body functions in many ways, even in the brain. The investigators are examining a possible role of bacteria of the nose and gut in the pathogenesis of PD. This may lead to a better understanding of what PD causes and may open new possibilities for diagnosis and treatment.

The investigators will recruit 100 PD patients and 100 control subjects. The investigators will characterize all subjects carefully with respect to clinical symptoms. The investigators will collect bacterial samples from the nose, mouth and stool of these subjects. Using modern genomic techniques the investigators will read out the genetic code of all bacteria contained in these samples and will be able to identify which species of bacteria are present in the samples. Using complex cluster computing the investigators will compare the pattern of bacterial species between PD patients and controls and look for specific abnormalities in PD patients.

If the investigators can detect specific differences of bacterial communities between PD patients and controls this may point to a role of bacteria as a cause of PD. Since there are many ways to influence bacterial communities pharmacologically (antibiotics, probiotics) it will be possible to investigate whether these therapies could alleviate or even reverse PD symptoms. Furthermore, the investigators would be able to use these differences as a biomarker which would enable us to develop a quick screening test for bacterial samples that may reveal whether a person has PD or not.

By doing this study the investigators will learn whether bacteria play a role in the development of PD and whether the investigators can use them as a biomarker or therapeutic target. So hopefully the investigators will be able in the future to better understand what causes PD, how the investigators can diagnose it as early as possible and how to cure patients from PD.

ELIGIBILITY:
Inclusion Criteria:

* over 50 years of age

Exclusion Criteria:

* Active smoking
* relevant gastrointestinal or ENT disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospital patients in- and outpatient From the community
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2011-11; Primary Completion 2015-04 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Filip Scheperjans, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (5):
- Finland (5):
  - Jorvi Hospital, Espoo
  - Helsinki University Central Hospital, Helsinki
  - Institute of Biotechnology, Helsinki University, Helsinki
  - Hyvinkää Hospital, Hyvinkää
  - Peijas Hospital, Vantaa